CLINICAL TRIAL: NCT03179865
Title: Evaluation of PUCAI Score at Assessment for Mucosal Healing During Clinical Remission in Pediatric Ulcerative Colitis
Brief Title: Evaluation of Early Mucosal Healing During Clinical Remission in Pediatric Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition unit, Wolfson Medical Center
Other Study IDs: 0114-16-WOMC
Record Dates: First submitted 2017-04-24; First posted 2017-06-07 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

SUMMARY:
Establishing that mucosal healing (MH) has occurred after therapy is an important treatment goal, and the gold standard is endoscopic evaluation. In UC it is unclear if clinical parameters are adequate. The pediatric ulcerative colitis activity index (PUCAI) has demonstrated good correlations for clinical remission and disease severity, but its role for establishing mucosal healing after therapy has not been validated . The ability to predict mucosal healing may be different for patients in long term remission compared to assessment after obtaining clinical remission. No previous study has prospectively validated the use of PUCAI as a proxy for MH specifically during clinical remission after therapy.

DETAILED DESCRIPTION:
All pediatric patients ≤ 19 years old and at the Wolfson Medical Center pediatric IBD center who enter clinical remission are routinely assessed by colposcopy or sigmoidoscopy assess. This is an analysis of prospectively collected data regarding PUCAI and endoscopic Mayo score at the time of assessment of mucosal healing by endoscopy. Patients could be included if they have establish ulcerative colitis, while they are on remission for at least 3 months after treatment of flare. For this study, complete clinical remission was absence of abdominal pain, and no diarrhea or bleeding (PUCAI<10). sigmoidoscopy will be performed between 12-24 weeks after remission was documented.

ELIGIBILITY:
Inclusion Criteria:

1. Ulcerative Colitis patient
2. clinical remission (PUCAI<10) for at least 3 months.
3. Sigmoidoscopy for assessment mucusa healing after therapy performed between 12-24 weeks after remission was documented

   -

   -

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients could be included if they have establish ulcerative colitis, while they are on clinical remission
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Mucusa healing according to the MAYO score | cross sectional study, the data will be reported during 4 years
  present of endoscopic disease defined by mayo score

CONTACTS AND LOCATIONS:
Locations (1):
- The Wolfson Medical Center, Holon, Israel